CLINICAL TRIAL: NCT01802645
Title: Open, Randomized, Multicenter Phase II Trial With Cetuximab /5-FU/FA/Irinotecan or Cetuximab/5-FU/FA /Irinotecan/Oxaliplatin in K-ras/B-raf Wild Type Patients or With Irinotecan/Oxaliplatin/5-FU/FA With or Without Bevacizumab in K-ras Mutant Patients as Neoadjuvant Treatment in Patients With Non- Resectable Colorectal Liver Metastases.
Brief Title: Cetuximab/FOLFIRI With or Without Oxaliplatin and FOLFOXIRI With or Without Bevacizumab in Neoadjuvant Treatment of Non-resectable Colorectal Liver Metastases
Acronym: CELIM2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-CELIM2-050; 2011-003288-31 (EudraCT Number)
Record Dates: First submitted 2013-02-11; First posted 2013-03-01 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: neoadjuvant; cetuximab; irinotecan; bevacizumab; oxaliplatin; 5-FU; Resection; colorectal liver metastases; liver resection; Chemotherapy; k-ras; non-resectable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab; Irinotecan; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cetuximab/FOLFIRI (Active Comparator): Cetuximab 250 mg/m² (1 h) weekly Irinotecan 180 mg/m² (1 h)*, d-l Folinic acid 400 mg/m² (2 h), 5-FU 400 mg/m² (Bolus), 5-FU 2400 mg/m² (46 h) every 2 weeks
  *reduced in UGT1A1 7/7 patients
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: 5-FU; Drug: Folinic Acid
- Cetuximab/FOLFOXIRI (Experimental): Cetuximab 250 mg/m² (1 h) weekly Irinotecan 125 mg/m² (1 h),* Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks
  *reduced in UGT1A1 7/7 patients
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-FU; Drug: Folinic Acid
- FOLFOXIRI (Active Comparator): Irinotecan 165 mg/m² (1 h)*, Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks
  *reduced in UGT1A1 7/7 patients
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-FU; Drug: Folinic Acid
- Bevacizumab/FOLFOXIRI (Experimental): Bevacizumab 5 mg/kg (30-90 min i.v.), Irinotecan 165 mg/m² (1 h),* Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks
  *reduced in UGT1A1 7/7 patients
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-FU; Drug: Folinic Acid

INTERVENTIONS:
Drug: Cetuximab
  Other Names: Erbitux
  Arms: Cetuximab/FOLFIRI; Cetuximab/FOLFOXIRI
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Bevacizumab/FOLFOXIRI
Drug: Irinotecan
  Other Names: Campto
Drug: Oxaliplatin
  Other Names: Eloxatin
  Arms: Bevacizumab/FOLFOXIRI; Cetuximab/FOLFOXIRI; FOLFOXIRI
Drug: 5-FU
  Other Names: 5-Fluorouracil
Drug: Folinic Acid
  Other Names: Leukovorin

SUMMARY:
The aim of this study is to investigate the following schedules for efficacy with regard to response rate in neoadjuvant treatment of patients with non-resectable liver metastases:

* Cetuximab/FOLFOXIRI and cetuximab/FOLFIRI in patients with ras wild type tumours and
* Bevacizumab/FOLFOXIRI and FOLFOXIRI in patients with ras mutant tumours.

DETAILED DESCRIPTION:
Patients with liver metastases from colorectal and without known extrahepatic metastases will be screened for this study including ras status (b-raf status according to local standard).

Patients receive chemotherapy according to the allocation and are re-evaluated for resectability every 8 weeks for a maximum of 6 months. Resectable patients will be resected and receive an adjuvant treatment to complete 12 cycles.

In certain circumstances, a second resection is allowed within the study.

Patients will be randomized using a web-based computer system that allows randomization if the key basic characteristics are entered.

Patients with ras wild-type tumours will be randomized to receive:

* Cetuximab/FOLFIRI or
* Cetuximab/FOLFOXIRI

Patients with ras mutations will be randomized to receive:

* FOLFOXIRI or
* FOLFOXIRI/bevacizumab

Chemotherapy doses are adjusted to the risk of toxicity in all treatment arms.

Stratification will be performed according to:

* Number of metastases (< 5 vs. ≥ 5 metastases)
* Primary tumour in situ
* Centre

Treatment regimens For dose reductions and conditions to continue please refer to the full protocol.

All drugs are used within the label and approved doses.

B-raf mutations are determined according to local standard. If a b-raf mutation is known before randomization, the investigator can consider the patient as ras wildtype OR as ras mutant patient.

Cetuximab/FOLFIRI :

Cetuximab 400 mg/m² (first dose, 2 h), then 250 mg/m² (1 h) weekly Irinotecan 180 mg/m², d-l Folinic acid 400 mg/m² (2 h), 5-FU 400 mg/m² (Bolus), 5-FU 2400 mg/m² (46 h) every 2 weeks

Cetuximab/FOLFOXIRI:

Cetuximab 400 mg/m² (first dose, 2 h), then 250 mg/m² (1 h) weekly Irinotecan 125 mg/m² , Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks

FOLFOXIRI:

Irinotecan 165 mg/m², Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks

Bevacizumab/FOLFOXIRI:

Bevacizumab 5 mg/kg (90 - 30 min i.v.), Irinotecan 165 mg/m², Oxaliplatin 85 mg/m² (2 h), d-l Folinic acid 400 mg/m² (2 h), 5-FU 3200 mg/m² (46 h) every 2 weeks

Evaluation for response and resections Patients are evaluated for response by the same imaging technique as at baseline every 8 weeks. The findings will be discussed for resectability within two weeks after tumour assessment in a local multidisciplinary team.

Technically resectable patients should be offered liver resection. The treatment will continue until liver resection or for a maximum of six months (12 cycles).

Adjuvant treatment After liver resection, an adjuvant treatment is recommended with the same schedule as preoperatively, for a maximum combined pre- and postoperative treatment of 12 cycles. If less than three postoperative cycles remain, no postoperative treatment will be started (see chapter 9.10).

Follow up After resection, patients will be followed up for 5 years after randomization. This includes

* imaging and clinical investigation every three months for the first 2 years, then every six months (patients without tumour progression / recurrence)
* survival status and surgical/medical treatment every three months for the first 2 years and then every six months (all patients)

ELIGIBILITY:
Patients can be enrolled, if all of these conditions apply:

1. Non-resectable, histologically confirmed, synchronous or metachronous colorectal liver metastases.
2. Non-resectability will be documented by a local multidisciplinary tumour board with participation of a surgeon experienced in liver surgery. Patients can be enrolled if they

   a) are technically non-resectable (locally determined by a multi-disciplinary team discussion based on remaining functional liver tissue after resection, i.e. i) involvement of both portal veins, all hepatic veins, portal vein of the liver lobe and hepatic veins draining the segments of the other liver lobe, or ii) other reasons for less than 30% remaining functional liver tissue after resection) and / or b) have ≥ 5 liver metastases and / or c) are regarded as non-resectable for other reasons (description necessary)
3. Patients with simultaneous liver metastases are eligible,

   1. if the primary tumour was resected at least 1 month prior to chemotherapy or
   2. all of the following conditions apply:

   i) the primary tumour is clearly resectable, ii) no radiation therapy is planned, iii) liver resection is planned before resection of the primary or at the same operation as the resection of the primary, iv) no two-stage liver resection is planned, and v) all efforts were made to exclude additional distant metastases.
4. WHO PS ≤ 1
5. Written informed consent
6. Adequate bone marrow function, liver function (neutrophils > 1.5 x 109/l; platelets > 100 x 109/l; haemoglobin > 5.0 mmol/l (8.0 g/dl); bilirubin ≤ ULN or ≤ 1.5 x ULN and not increasing more than 25 % within the last 4 weeks; SGOT and SGPT < 5 x UNL)
7. Age ≥ 18 years

Exclusion Criteria:

1. Any evidence of extrahepatic metastases, distant lymph node metastases and primary tumour recurrence
2. (deleted)
3. Prior systemic anti-tumour therapy with anti- EGFR-, anti-angiogenetic drugs or with chemotherapy (except adjuvant chemotherapy with an interval of ≥ 6 months or in combination with radiation as radio sensitizer)
4. Radiotherapy or major abdominal or thoracic surgery (excluding diagnostic interventions or venous port implantation) ≤ 4 weeks before study entry
5. Renal insufficiency with serum creatinine ≥ 1.5 x UNL. If serum creatinine is between 1.0 and 1.5 x UNL, the creatinine clearance according to the Cockroft-Gault formula should be ≥ 60 ml/min
6. Hypertension with an arterial blood pressure > 150/90 mmHg
7. Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last 12 months, significant arrhythmias)
8. Known proteinuria > 1 g/day (to be tested if proteinuria more than 1+ in the urinary dipstick analysis)
9. Peripheral neuropathy > CTC grade I
10. Concurrent systemic immune therapy, chemotherapy, hormone therapy, or patients receiving immune suppressive treatment (i.e. for transplantation, severe rheumatologic disease)
11. Participation in clinical trials with investigational agents within 30 days before start of the treatment in study
12. Active treatment of

    1. peptic ulcers or bleeding erosive esophagitis / gastritis within 3 months before study
    2. pulmonary embolism, severe or unstable angina pectoris or myocardial infarction, stroke or transient ischemic attack within 12 months before study
    3. deep vein thrombosis within 4 weeks before study
13. Inflammatory bowel disease
14. History of other malignancies, from which the patient is not 5 years disease free, with the exception of colorectal cancer, or adequately treated basal cell or squamous cell carcinoma of skin or in-situ cervical cancer within 5 years before study
15. History of brain metastases
16. History of severe psychiatric illness
17. Active drug- or alcohol abuse
18. Known hepatitis B or C or HIV infection
19. Breast- feeding or pregnant women
20. Lack of effective contraception (for male and female patients)
21. Known intolerance to one of the following drugs: cetuximab, bevacizumab, oxaliplatin, irinotecan, 5-FU, folinic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | up to 1 year after randomization
  Rate of patients with partial or complete response according to modified RECIST criteria.

SECONDARY OUTCOMES:
Rate of resected patients without early relaps | 6 months after resection
  Rate of patients who had a R0 resection of all lesions and are disease free for at least 6 months in the ITT population.

OTHER OUTCOMES:
R0 resection rate | up to 1 year after randomization
  Resection rate, defined as patients with microscopically complete (R0) resection (ITT- population)
Resection rate | up to 1 year after randomization
  Rate of liver resection with macroscopically tumour free margins and/or RFA (all patients with R0 or R1 resection and/or complete RFA of all lesion, ITT- population)
Progression free survival | up to 3 years after randomization
  Progression free survival (Medium, Kaplan-Meier-estimation, ITT- population)
Disease free survival after resection | up to 3 years after resection
  Disease free survival after resection (Medium, Kaplan-Meier-estimation, resected patients)
Overall survival | up to 5 year after randomization
  Overall survival (Kaplan-Meier-estimation, ITT- population)
Toxicity | up to 1 year after randomization
  Toxicity according to NCI-CTC criteria v. 4.0 Perioperative toxicity according to Clavien
Pathological response | up to 1 year after randomization
  Pathological response in the resected tumour tissue
Molecular markers | up to 1 year after randomization
  Evaluation of molecular predictive markers for response (i.e. other mutations in EGFR signalling pathway, EGFR ligands) and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Folprecht, PD Dr., Principal Investigator — University hospital "Carl Gustav Carus" Dresden
Locations (15):
- Germany (15):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Charité Campus Virchow, Berlin
  - Überörtliche Gemeinschaftspraxis Hämatologie/ Onkologie, Bocholt
  - Klinikum Coburg GmbH, Coburg
  - Onkologie Dülmen GbR, Coesfeld
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Klinikum der Johann Wolfgang Goethe Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Landshut gGmbH, Landshut
  - University hospital Leipzig, Leipzig
  - Johannes-Gutenberg-Universität, Mainz
  - Klinikum Oldenburg GmbH, Oldenburg
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Universitätsklinikum Würzburg, Würzburg